CLINICAL TRIAL: NCT04072601
Title: Statins for Prevention of Disease Progression and Hospitalization in Liver Cirrhosis: A Multi-center, Randomized, Double Blind, Placebo-controlled Trial. The STATLiver Trial
Brief Title: Statins for Prevention of Disease Progression and Hospitalization in Liver Cirrhosis
Acronym: STATLiver
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study part one completed
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: University of Copenhagen (Other); Aarhus University Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nina Kimer, MD, PhD, Clinician Researcher, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STATLiver2019
Record Dates: First submitted 2019-06-05; First posted 2019-08-28 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Liver Cirrhoses
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Part One: Enrolment of 48 participants. Evaluation of safety, resources and recruitment.
  If adequate, Part Two: Enrolment up to 162 participants.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation and randomisation is blinded. Participants are only identified by randomisation number (no group names) Allocation ratio is 1:1 All personnel and participants are blinded through the study period. All outcome assessors are blinded to treatment, and initial data analysis is performed blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atorvastatin (Experimental): Atorvastatin 10-20 mg for 18 months of treatment. Start dose is 10 mg, adjusted to 20 mg after 15-30 days if no sideeffects occurs.
  Interventions: Drug: Atorvastatin 10mg
- Control (Placebo Comparator): Placebo of atorvastatin 10 mg, 1-2 tablets for 18 months of treatment. Start dose is 1 tablet (10 mg placebo), adjusted to 2 tablets (20 mg placebo) after 15-30 days if no side effects occurs.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Placebo oral tablet — Lactose monohydrate 50 mg, potato starch 45 mg, Gelatine 1,2 mg, Magnesium stearate 0,5, Talc 4,5 mg
  Arms: Control
Drug: Atorvastatin 10mg — Tablet, can be adjusted to 2 tablets if tolerated
  Arms: Atorvastatin

SUMMARY:
In a randomized, doubleblind and placebo-controlled trial we assess both clinical and cellular effects of atorvastatin in patients with liver cirrhosis.

162 participants will be allocated to atorvastatin 10-20 mg or placebo for 18 months. Clinical outcomes of survival, hospitalizations and safety will be evaluated. Also, the trial will investigate cellular functions in the liver by mass spectrometry proteomics, and single cell transcriptomics as well as exploring atorvastatin effects on different fenotypes by metagenomics.

DETAILED DESCRIPTION:
Introduction Several studies have demonstrated the beneficial effects of statins in vascular and heart disease. Statins have antithrombotic effects, decrease oxidative stress and inflammation at the vessel wall, and improve endothelial dysfunction by increasing Nitric Oxide (NO) production in endothelial cells.

Statins may also inhibit fibrogenesis in cirrhotic rats. In recent years, a series of pilot studies have assessed the effects of simvastatin on portal hypertension and risk of variceal bleeding.

Only a few studies have evaluated the efficacy of statins in cirrhosis of mixed etiology and decompensated cirrhosis. High quality clinical trials have focused on the hemodynamic effects of simvastatin on portal hypertension. Evidence supporting the use of statins in a real-world clinical setting, and data on the effects on inflammation and generation of fibrosis in the liver in humans is in high demand.

Study setting The trial will take place in university hospitals with tertiary referral from other hospitals, departments and general practice. Patients referred to the outpatient clinics or hospitalized in the Gastro Unit, Amager Hvidovre Hospital (AHH) and Department of Hepatology and Gastroenterology, Aarhus University Hospital (AUH), all Denmark are eligible for inclusion.

Study Part One

After enrolment of the first 48 participants an evaluation of the trial feasibility will performed on the following parameters:

i) recruitment rates, ii) allocation of adequate resources to the trial, iii) safety for the participants.

Study Part One will deliver data to conduct a pilot study on the exploratory endpoints of inflammation, proteomics and metabolomics.

The substudy will apply the following methodology:

Initial analyses of biological material are performed blinded based on studyID, without revealing allocation to atorvastatin or placebo.

Comparison between groups are performed by blinded allocation, meaning that analysis are performed as: group A versus group B, without prior knowledge of which group received the active drug.

Scientific evaluation and clinical translation of study results and data are only performed after revelation of which group received the active drug.

Study Part Two

If the steering committee find all three conditions: recruitment, resources and safety adequate, the trial will continue into Part Two, with enrolment up to 162 participants as required to balance the clinical endpoints.

Criteria for discontinuation of intervention:

Discontinuation of trial drug will be performed in case of:

* The participant withdraws informed consent.
* Participants reach a primary endpoint (death or liver transplantation).
* The participant experiences serious adverse events that cause a risk to the participant's life or viability.
* The participant develops toxicity, intolerance or allergy associated with intervention medication.
* The trial participant is admitted to hospital for other morbidity that is incompatible with further treatment with atorvastatin.
* Blinding is revealed.
* A trial participant will be classified as dropped out of the study if the participant has ingested less than 55 % of atorvastatin or placebo at days 180.

Statistical methods Data will be analyzed as repeated measures Analysis of variance (ANOVA). Independent groups will be compared using unpaired T-test or non-parametric tests depending on normality distribution of data. Survival analysis will be performed by Cox-regression analyses.

Statistical analyses will be performed as per protocol and as intention to treat analyses.

Missing data will not be replaced but left blank in statistical analysis. For intention to treat analyses on repeated measures, the last available value will be carried forward to last value.

Sample Size

Prior data may indicate that the median survival time on the control treatment is 35 months. If the true hazard ratio (relative risk) of control subjects relative to experimental subjects is 0.52, we will need to study 70 experimental subjects and 70 control subjects to reject the null hypothesis that the experimental and control survival curves are equal with probability (power) 0.85. The Type I error probability associated with the test of this null hypothesis is 0.05.

With an expected drop-out rate of fifteen percent, we plan to enroll in total 162 participants in Study Part One and Two, to reach the clinical endpoint of survival.

Auditing The trial will be approved by the Danish Authorities of Health and Medicine, and may be subject to auditing by this institution, independent of the sponsor and investigators. Investigator allows direct access to source data and documents (including patient records) used in the trial for monitoring, auditing and/or inspection from GCP-units and The Danish Medicines Agency.

Bio bank A biobank containing blood and liver tissue is established for the trial. The bio bank contains both samples for planned analyses, and in case of excess material, samples will be stored in a bio bank for future research.

All investigations and results derived from the bio bank for future research will serve the purpose of improving the life and health of patients with liver cirrhosis.

Research ethics approval Registration by the Danish Data protection Agency was conducted April 9, 2019. Application for approval at the Scientific Ethics Committees of the Capital Region of Denmark was approved by: September 3, 2019, with ammendments approved by: January 20, 2020 (protocol version 2) and August 7, 2020 (protocol verison 3).

Legal assistance Legal advice for contracts and agreements is provided by Centre for Innovation and Research, The Capital Region of Denmark c/o Cobis, Ole Maaløes vej 3, DK-2200 Copenhagen N.

Declaration of interests Authors of this protocol have no financial interests (holds no stakes, no ownership, and do not provide academic services) to any medical companies involved in producing or marketing statins.

Insurance Patients participating in this trial will be insured through the national patient insurance. Trial participants are informed of this relation in written information of trial participant's rights. Sponsor and investigators are covered by statutory insurance from AHH and AUH.

Dissemination policy This study will support an open access policy and aims to prepare all collected data to publication in anonymized form in an open access database after dissemination of the pre-defined trial outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age of 18 to 80 years
* Patients with liver cirrhosis, diagnosed by liver biopsy or ultrasound or CT scan of the liver and clinical biochemistry compatible with cirrhosis within the past 3 months.
* In women, documented absence of pregnancy and unless in menopause commitment to use adequate contraception.
* Clinically significant portal hypertension with a hepatic venous pressure gradient measured by liver vein catheterization >10 mmHg.
* Ability to read and understand project information in Danish and give written, informed consent.

Exclusion Criteria:

* People treated with statins within the last year.
* People with liver cirrhosis, with a clinically verified infection (standard biochemistry, culture) within the last four weeks.
* Pregnancy or lactation.
* Hepatocellular carcinoma
* HIV infection and treatment with protease inhibitors
* People in whom the clinician and investigators may have reason to doubt compliance to trial medication
* Clinical and biochemical signs of hepato-renal syndrome defined by current guidelines (EASL) within the last 14 days
* A MELD score above 23, or Child-Pugh score higher than 13.
* Hepatic encephalopathy grade 2 or higher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of numbers of death or liver transplantation | 1.5 years
Number of hospitalizations with liver related complications | 1.5 years

SECONDARY OUTCOMES:
Number of adverse events | 1.5 years (18 months)
Number of Patients developing decompensation of liver cirrhosis | 1.5 and 5 years
Inflammation and macrophage activation | 0.5 and 1.5 years
  Markers of systemic inflammation (TNF-alfa, IL4, IL10, IL 18, hsCRP) and macrophage activation (CD163, surface Mannose receptor) is measured before and after intervention
Change in clinical score | 0.5, 1.5 years
  MELD score a calculated score including parameters of bilirubin, INR, and creatinin levels. The score is calculated using log values. Range 5->30, with a higher score indicating worse outcome for patients.
Numbers of episodes of decompensation | 1.5 and 5 years
Change in clinical score Child-Turcotte-Pugh | 0.5 and 1.5 years
  Child score, a sum of point given on five parameters: P-albumin, P-bilirubin, Coagulation factor II,VII,X; presence of ascites and presence of hepatic encephalopathy. Score range: 5-15 with high score predicting af worse outcome
Protein activity in the hepatic stellate cell | 0.5 years
  By high-sensitivity Mass spectrometry-based proteomics, we will perform proteomics analysis of hepatic stellate cells and Kupffer cells under atorvastatin influence
Cell activation | 0.5 years
  Gene activation by transcriptomics of mRNA in the hepatic stellate cell, combined with protein activity by mass spectrometry proteomics
Change in clinical score | 0.5, 1.5 years
  Short Physical performance battery, a combined score of three physical tests, chair.-stand, gait speed and balance. Range 0-12 points, a high score indicates better physical performance.
Time to first hospital admission due to decompensation or complications of liver cirrhosis | 1.5 and 5 years
Patient survival | 1.5 and 5 years
Composite endpoint of numbers of death or liver transplantation | 5 years
Number of hospitalization with liver related complications | 5 years
Change in clinical score, Frailty Index | 0.5, 1.5 years
  Frailty Index, a questionnaire based on patients selfperceived health and performance. This score is under development and validation during this and other trials.

CONTACTS AND LOCATIONS:
Overall Officials: Thit M Kronborg, MD, Principal Investigator — Gastro Unit, Hvidovre University Hospital; Flemming Bendtsen, DmSci, Study Chair — Gastro Unit, Hvidovre University Hospital
Locations (1):
- Gastro Unit, medical Division, University Hospital Hvidovre, Hvidovre, Danmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
IPD and supporting information are planned to be shared via data repository sites, such as UCPH data repository or other public data repository.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be stored for up to 10 years after completion of the trial, depending on approval from Danish Health Authorities, Scientific Ethics Comittee and the Danish Data Protection Regulation.
Access Criteria: upon request

REFERENCES:
- [Background] Lefer DJ. Statins as potent antiinflammatory drugs. Circulation. 2002 Oct 15;106(16):2041-2. doi: 10.1161/01.cir.0000033635.42612.88. No abstract available. PMID 12379569
- [Background] McGirt MJ, Lynch JR, Parra A, Sheng H, Pearlstein RD, Laskowitz DT, Pelligrino DA, Warner DS. Simvastatin increases endothelial nitric oxide synthase and ameliorates cerebral vasospasm resulting from subarachnoid hemorrhage. Stroke. 2002 Dec;33(12):2950-6. doi: 10.1161/01.str.0000038986.68044.39. PMID 12468796
- [Background] Chong LW, Hsu YC, Lee TF, Lin Y, Chiu YT, Yang KC, Wu JC, Huang YT. Fluvastatin attenuates hepatic steatosis-induced fibrogenesis in rats through inhibiting paracrine effect of hepatocyte on hepatic stellate cells. BMC Gastroenterol. 2015 Feb 15;15:22. doi: 10.1186/s12876-015-0248-8. PMID 25886887
- [Background] Zafra C, Abraldes JG, Turnes J, Berzigotti A, Fernandez M, Garca-Pagan JC, Rodes J, Bosch J. Simvastatin enhances hepatic nitric oxide production and decreases the hepatic vascular tone in patients with cirrhosis. Gastroenterology. 2004 Mar;126(3):749-55. doi: 10.1053/j.gastro.2003.12.007. PMID 14988829
- [Background] Abraldes JG, Albillos A, Banares R, Turnes J, Gonzalez R, Garcia-Pagan JC, Bosch J. Simvastatin lowers portal pressure in patients with cirrhosis and portal hypertension: a randomized controlled trial. Gastroenterology. 2009 May;136(5):1651-8. doi: 10.1053/j.gastro.2009.01.043. Epub 2009 Jan 24. PMID 19208350
- [Background] Cash WJ, O'Neill S, O'Donnell ME, McCance DR, Young IS, McEneny J, McDougall NI, Callender ME. Randomized controlled trial assessing the effect of simvastatin in primary biliary cirrhosis. Liver Int. 2013 Sep;33(8):1166-74. doi: 10.1111/liv.12191. Epub 2013 May 15. PMID 23672463
- [Background] Pollo-Flores P, Soldan M, Santos UC, Kunz DG, Mattos DE, da Silva AC, Marchiori RC, Rezende GF. Three months of simvastatin therapy vs. placebo for severe portal hypertension in cirrhosis: A randomized controlled trial. Dig Liver Dis. 2015 Nov;47(11):957-63. doi: 10.1016/j.dld.2015.07.156. Epub 2015 Aug 6. PMID 26321186
- [Background] Abraldes JG, Villanueva C, Aracil C, Turnes J, Hernandez-Guerra M, Genesca J, Rodriguez M, Castellote J, Garcia-Pagan JC, Torres F, Calleja JL, Albillos A, Bosch J; BLEPS Study Group. Addition of Simvastatin to Standard Therapy for the Prevention of Variceal Rebleeding Does Not Reduce Rebleeding but Increases Survival in Patients With Cirrhosis. Gastroenterology. 2016 May;150(5):1160-1170.e3. doi: 10.1053/j.gastro.2016.01.004. Epub 2016 Jan 14. PMID 26774179
- [Result] Kalinowski L, Dobrucki LW, Brovkovych V, Malinski T. Increased nitric oxide bioavailability in endothelial cells contributes to the pleiotropic effect of cerivastatin. Circulation. 2002 Feb 26;105(8):933-8. doi: 10.1161/hc0802.104283. PMID 11864921
- [Derived] Kimer N, Gronbaek H, Fred RG, Hansen T, Deshmukh AS, Mann M, Bendtsen F. Atorvastatin for prevention of disease progression and hospitalisation in liver cirrhosis: protocol for a randomised, double-blind, placebo-controlled trial. BMJ Open. 2020 Jan 23;10(1):e035284. doi: 10.1136/bmjopen-2019-035284. PMID 31980514
- See also: @Nkimer is a twitter account posting progress on the StatLiver trial — https://twitter.com/NKimer